CLINICAL TRIAL: NCT02293889
Title: The Impact of Physical Activity and Vitamin D on Osteoarthritic Knee Pain in Older Obese People
Brief Title: Impact of Physical Activity and Vitamin D on Osteoarthritic Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NO 188
Record Dates: First submitted 2014-11-13; First posted 2014-11-19 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Pain; Vitamin D; Physical activity; Pilot study; Qualitative Interview; Obesity; Older adults
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Motor Activity; Obesity | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vitamin D (Experimental): Vitamin D3 2000IU/daily 3 months
  Interventions: Dietary Supplement: Vitamin D3 2000IU/daily 3 months
- Physical Activity (Experimental): PA intervention People with Osteoarthritis Walking Programme
  Interventions: Behavioral: PA intervention People with Osteoarthritis Walking Programme
- Vitamin D and Physical Activity (Experimental): Vitamin D3 2000IU/daily 3 months PA intervention People with Osteoarthritis Walking Programme
  Interventions: Dietary Supplement: Vitamin D3 2000IU/daily 3 months; Behavioral: PA intervention People with Osteoarthritis Walking Programme
- Placebo (Placebo Comparator): Placebo capsule: edible oil
  Interventions: Other: Placebo capsule (Vitamin D): edible oil

INTERVENTIONS:
Dietary Supplement: Vitamin D3 2000IU/daily 3 months — Vitamin D will be provided in the form of a daily capsule over 3 months containing 2000IU of Vitamin D3 suspended in oil (manufactured and provided by DSM) with the aim of raising 25OHD levels to sufficiency (>50nmol/L) by 3 months.
  Arms: Vitamin D; Vitamin D and Physical Activity
Behavioral: PA intervention People with Osteoarthritis Walking Programme — The PA intervention will aim to increase levels of PA safely in our defined population. Participant are given a pedometer at the start of the intervention and encouraged to record their daily step counts and set step goals using the online system provided (POW: People with osteoarthritis walking programme).
  Arms: Physical Activity; Vitamin D and Physical Activity
Other: Placebo capsule (Vitamin D): edible oil — Placebo capsules will be administered over 3 months, as daily capsules (identical to Vitamin D capsules) containing edible oil (manufactured and provided by DSM)
  Arms: Placebo

SUMMARY:
Knee Osteoarthritis (KOA) is a major cause of pain and disability, particularly in those of increasing age and body fat. As there are no very effective therapies for KOA, disease often progresses until knee replacement surgery is needed. It has been observed Vitamin D and Physical Activity (PA) levels are lower in those with KOA, increased age and body fat. As the relationship between KOA, Vitamin D and PA levels are not clearly understood, this study aims to explore these relationships and the acceptability/feasibility of PA and Vitamin D interventions in those who would likely to benefit from these interventions.

200-300 people, 50-70 years, BMI 30-40kg/m2, meeting American College of Rheumatology (ACR) KOA Guidelines, will be recruited from North Tyneside and Liverpool Hospital trusts November 2014-January 2016 to participate in a single cross-sectional study visit, which will measure: Vitamin D/Calcium serum levels, BMI/Body Fat, mobility, Quality of life and pain (by questionnaire), and PA levels.

Those participants with insufficient Vitamin D levels (25-50nmol/L) and PA levels (<30min moderate PA/week), will be invited to take part in a 3 month pilot RCT study.

>64 people will be recruited for the pilot RCT and equally randomly allocated to 1 of 4 intervention groups: Vitamin D (1 capsule a day: 2000IU), Placebo (identical capsule: 1 a day), PA (online PA programme) and PA and Vitamin D. Additionally at the end of the 12 week study visit, up to 20 participants will be invited to take part in a qualitative interview exploring their experience during the two studies.

DETAILED DESCRIPTION:
The primary aim of this project is to test the feasibility and acceptability of increasing PA and Vitamin D supplementation interventions in older, obese people with knee osteoarthritis, with low baseline levels of PA and Vitamin D by performing a 2*2 design pilot randomized controlled trial and a qualitative interview.

The secondary aims of this project is to:

1. Explore the relationships between Vitamin D levels, PA levels and KOA pain (using cross-sectional study results)
2. Estimate effect sizes and inter-individual variation which can be used in the design of a future definitive RCT.

The project refers to 2 integrated studies:

* Firstly a cross-sectional study to identify individuals with low vitamin D concentrations, low Physical activity levels, who are obese and who meet the ACR KOA criteria for knee osteoarthritis.
* Secondly a pilot randomized controlled trial, which aims to test the feasibility and acceptability of administering vitamin D or placebo capsules and increasing physical activity over a 3 month period.

These 2 studies will run consecutively over 2 winter periods or phases: phase 1 (November 2014- January 2015: cross sectional study followed by intervention study (February 2015- May 2015). Phase 2 will run over the same time periods 1 year later.

1. Cross-sectional study potential participant identification (November 2014-January 2015):

   On Tyneside, the investigators will identify potential participants by screening GP surgery patient lists against inclusion criteria (see A17-1). At the Liverpool site, participants will be identified by research staff at hospital clinics (obesity). Potentially eligible people will be mailed/given a letter of invitation, together with information about the study and a consent form to take home and consider. Those interested in joining the study will be invited to contact their local research team using the contact information provided.
2. Cross-sectional study screening(November-January 2014/15):

   Potential participants will complete a brief telephone screening questionnaire when they call to register their interest in the study to verify their eligibility. The CI will then call back to inform the potential participant of their eligibility and, if eligible, an appointment will be made to attend for the cross-sectional study visit (study visit 1).
3. Cross-sectional study visit: study visit 1 (November-January 2014/15):

   Participants will attend an appointment at North Tyneside General Hospital or Aintree Hospital Liverpool (depending on their research site) lasting 1 hour 30 minutes. The visit will begin by reviewing the participant information sheet and completing the consent form. After this, several measurements will be completed:
   * Blood samples
   * Questionnaires
   * Body composition At the end of the study visit, the participants will be given a accelerometer to wear for the next 3 days. Participants will be provided with instructions on accelerometer use, activity log and a prepaid envelope in which to return the device.
4. Screening for eligibility for pilot RCT (January 2015):

   Using data from the cross-sectional study, participants with low vitamin D concentration (25-50nmol/L) and low physical activity levels (<30min/week moderate activity)will be invited to participate in the pilot RCT.
5. Pilot RCT starter session (study visit 2) (February 2015/16):

   Participants will attend a starter session for the pilot RCT study at North Tyneside General Hospital or Aintree hospital Liverpool. Prior to their appointment, all participants will be randomly allocated (stratified by gender) to 1 of 4 treatment arms:
   * Vitamin D supplementation: 2000IU/day vitamin D capsule
   * Placebo: 1/day edible oil capsule (identical to vitamin D capsule)
   * Physical activity intervention (online system to record daily step using a pedometer provided, which slowly increase step and physical activity goals)
   * Vitamin D + Physical activity intervention.

   The investigator will explain how to undertake the intervention, provide study materials and answer any questions the participant may have. Vitamin D and Placebo intervention will be blinded to the participants.
6. 6 week follow up (study visit 3)(March 2015/16: All pilot RCT participants will be invited back at 6 weeks into their intervention period for a study visit lasting 1-1hr 15 minutes, at either NTGH or UHA. The same measurements taken during the cross-sectional study visit will be taken with some additional compliance measures.
7. 12 week follow up (study visit 4) (April/May 2015/16): All pilot RCT participants will be invited back at 12 weeks into their intervention period for a study visit lasting 1-1hr 15 minutes at NTGH or UHA. This will be the study close for those not taking part in the qualitative interview. The same measurements will be taken as in study visit 3. Participants will be mailed feedback on their study measures including vitamin D status.
8. Qualitative interview (April/May 2015/16):

A subset of up to 20 participants will be invited to take part in a qualitative interview at NTGH or UHA directly after study visit 4. The interview will last 1hr and explore participants views in a range of topics which may identify areas of improvement in the design, delivery or practical arrangements of the studies in order to inform future studies in this area.

ELIGIBILITY:
Inclusion Criteria:

CROSS SECTIONAL STUDY

1. Obese: BMI 30-40kg/m2 as defined by WHO criteria
2. Older adults: 50 - 70 years
3. OA of the knee according to ACR Guidelines on symptomatic Knee OA criteria (using history and physical examination:

   • Pain in the knee

   AND 3 OF THE FOLLOWING:
   * Over 50 years of age
   * Less than 30 minutes of morning stiffness
   * Crepitus on active motion
   * Bony tenderness
   * Bony enlargement
   * No palpable warmth of synovial
4. Good understanding of written and spoken English (as no translation services will be available to this study).

PILOT STUDY

All of the inclusion criteria for the cross-sectional study (above), plus:

1. Low objectively measured levels of Vitamin D, defined as:

   Insufficient (25-50nmol/L), excluding deficient (<25 nmol/L), the 25OHD concentration at which symptoms as a result of Vitamin D deficiency commonly occur.
2. Low PA recorded from accelerometers defined as:

<30min/week of moderate PA, <15min/week vigorous PA (2*credit of moderate activity) defined as being 'inactive' by UK government guidelines. Activities only counted if they occurred in >10mins bouts. Activity was defined as moderate if it made the participant 'breathe faster, feel warmer or sweat' and increased heart rate. Activities identified as moderate included: brisk walking, cycling, gardening, housework, DIY, climbing stairs and carrying heavy loads.

Exclusion Criteria:

CROSS-SECTIONAL STUDY

1. Any other type of arthritic condition, e.g. RA, Fibromyalgia, Ankylosing Spondylitis, Gout, Lupus, Paget's Disease, Polymyalgia rheumatic (PMR), Psoriatic arthritis, Scleroderma, Sjogrens Syndrome
2. Currently taking part in a PA/exercise regime
3. Taking Vitamin D, cod liver oil or Calcium capsules/supplements (topical/oral/intravenous, prescribed/non-prescribed) above 10µg/day of vitamin D and/or 500µg/day of calcium.
4. Taking part in another intervention/trial (depending on researchers discretion)
5. Chronic alcohol abuse (> 21 (women) and 28 (men) SI units/week

PILOT STUDY

The same exclusion criteria as the cross-sectional study, plus:

1. Conditions which can interfere with Vitamin D supplement adsorption:

   * Malabsorption syndromes: e.g. cystic fibrosis, celiac disease, whipples disease, Crohns Disease, Bypass Surgery, short bowel syndrome,
   * Diagnosed restrictive eating disorder
   * Hypercalcaemia (albumin-adjusted plasma calcium > 2.60 mmol/l)
   * Hypocalcaemia (albumin-adjusted plasma calcium < 2.15 mmol/l)
   * Renal Stage 4-5 Chronic Kidney Disease: GFR < 30 ml/min/1.73m2
   * Primary hyperparathyroidism
2. Conditions which can affect normal baseline levels of vitamin D:

   * Current pregnancy, delivery of child/breast feeding 1 year prior to recruitment
   * Holiday with significant sunlight exposure (specified by list of sunny destinations) in the last 3 months and plans for holidays to sunny/skiing destinations for the duration of the study.
   * Current Anticonvulsant drug therapy
   * Current Glucocorticoid use
   * Current HIV/treatment with Antiretroviral drugs
   * Current anti-oestrogen (aromatase inhibitors, oestrogen receptor inhibitors and selective oestrogen receptor moderators) such as used to treat breast cancers
   * Those currently taking cytostatic/anti-tumour drugs
   * Granulomatous disorders: sarcoidosis, TB, Lymphomas
3. Current conditions which may be made worse/prompts complications of by vitamin D consumption

   * Chronic Renal Disease: stage 4 and 5 (see above)
   * Liver disease
   * Histoplasmosis
   * hyperparathyroidism
   * Hypocalcaemia or hypercalcemia (as defined above)
   * Lymphoma
   * Current/recent (in the last 6 months) supplementation(topical/oral/intravenous, prescribed and non-prescribed) with: Phosphorous, >10µg/day Vitamin D and >500mg/day Calcium

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of intervention by qualitative interview | 1 hour
  Qualitative interview with n=20 after last pilot RCT study visit. Interviews will be audio recorded, transcribed and analyzed using a thematic approach using NVivo software to identify main issues.

SECONDARY OUTCOMES:
Self reported knee joint pain and function by WOMAC Questionnaire | 15 mins
  Questionnaire designed to measure osteoarthritic pain specifically, administered at cross sectional and follow up pilot RCT study visits.
Objectively measured (by accelerometer) physical activity | 3 days
  PA will be measured after cross-sectional study visit and pilot RCT follow up visits.
Serum vitamin D concentrations measured by venous blood sample | 10 mins
  Venous blood samples taken at cross-sectional study visit and pilot RCT follow up visits, processed and serum sent to DSM for analysis.
Serum vitamin D concentrations measured by Dried Blood Spot sample | 10 mins
  Dried blood spot samples taken at cross-sectional study visit and pilot RCT follow up visits, processed and DBS cards sent to DSM for analysis.
Serum Calcium concentrations measured by venous blood sample | 10 mins
  Venous blood samples taken at cross-sectional study visit and pilot RCT follow up visits, processed and brought to Freeman Hospital Laboratory for analysis.
Musculoskeletal function measured by Timed up and go test | 15 mins
  Timed up and go test performed at cross-sectional study visit and pilot RCT follow up visits
Body composition measured by Tanita scales | 10 mins
  Weight, BMI and body Fat % measured using Tanita Bio impedance scales at cross-sectional study visit and pilot RCT follow up visits
Height measured by stadiometer | 5 mins
  Height in cm measured using stadiometer at cross-sectional study visit and pilot RCT follow up visits
Waist circumference measured using tape measure | 5 mins
  Waist circumference measured in cm at cross-sectional study visit and pilot RCT follow up visits
Quality of life measured using SF-36 Questionnaire | 10-15 mins
  Questionnaire specifically designed to measure physical and metal quality of life will be completed by participant at cross-sectional study visit and pilot RCT follow up visits

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Brown, MSc, Study Chair — Newcastle University; John C Mathers, PhD, Principal Investigator — Newcastle University
Locations (2):
- United Kingdom (2):
  - Aintree University Hospital, Liverpool
  - North Tyneside General Hospital, Newcastle upon Tyne